CLINICAL TRIAL: NCT03173911
Title: Effects of the Elastic Bandage on the Postural Balance of Young Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Norte do Paraná (Other)
Responsible Party: Principal Investigator, Helen Christofel, Master student, Universidade Norte do Paraná
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Projeto Kinesio
Record Dates: First submitted 2017-05-29; First posted 2017-06-02 (Actual); Last update posted 2017-06-02 (Actual); Status verified 2017-05

CONDITIONS: Postural Control
Keywords: Balance; Postural control; Elastic Bandages; Force plate
MeSH Terms: interventions — Bandages; Compression Bandages

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial where participants will be allocated into four intervention groups: G1 (n = 12) will receive therapeutic elastic bandage by the Therapy Taping® method (BET) in the ankles; G2 (n = 12) will receive the application of the BET in the lumbar region and G4 (n = 12) will receive the application for all the strategies. The individuals' balance will be evaluated in four moments: pre-intervention (Pre), immediately (Ime), 24 and 48 hours after intervention (24h and 48h). The main equilibrium parameters analyzed will be: ellipse area (95%) of COP in square centimeters (A-COP in cm2), average speed in centimeters per second (VM in cm / s) and average frequency in Hertz (FM in Hz) Of COP oscillations in the anterior-posterior (A / P) and mid-lateral (M / L) directions, during three postural control tasks: open-eye semitandem (STOA) and right and left unipodal support (UNPD And UNPE).
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (4):
- Ankle (Active Comparator): composed by 12 participants who will receive the application of the bandage for the ankle strategy in both lower limbs, being determined the application of the technique in I without fixed point, from medial malleolus to lateral malleolus passing under the hindfoot, finally a cleavage technique passing over the malleoli and ending in the anterior region of the ankle joint. The balance of each individual will be evaluated in the force platform at four different times, before, immediately after, after 24 and 48 hours after the application of the bandage, in three different tasks of postural control in the force platform, being: unipedal right, unipedal left and task Of bipedal support in the semi-tandem position. Will be performed three evaluations of 30s each, with 30s of interval between each evaluation.
  Interventions: Device: Bandage
- Hamstrings (Active Comparator): composed by 12 participants who will receive the application of the bandage for the posterior thigh (hamstrings) strategy in both lower limbs. The technique will be determined in I with fixed point of the skin of the ischial tuberosity and moving point until the Lateral tibia (near the head of the fibula) and medial tibia (goose-foot insertion). The balance of each individual will be evaluated in the force platform at four different times, before, immediately after, after 24 and 48 hours after the application of the bandage, in three different tasks of postural control in the force platform, being: unipedal right, unipedal left and task Of bipedal support in the semi-tandem position. Will be performed three evaluations of 30s each, with 30s of interval between each evaluation.
  Interventions: Device: Bandage
- Lumbar (Active Comparator): composed by 12 participants who will receive the application of the bandage for the hip (lumbar) strategy, being determined the application of the technique in I with fixed point in the ischial tuberosity and moving point until the height of the last ribs, making a cleavage in the Height of the superior iliac spine. The balance of each individual will be evaluated in the force platform at four different times, before, immediately after, after 24 and 48 hours after the application of the bandage, in three different tasks of postural control in the force platform, being: unipedal right, unipedal left and task Of bipedal support in the semi-tandem position. Will be performed three evaluations of 30s each, with 30s of interval between each evaluation.
  Interventions: Device: Bandage
- Total (Active Comparator): composed by 12 participants who will receive the application of the bandage for all strategies in both lower limbs, being determined the application of the technique in I with fixed point in the II and III toes and moving point until the height of the last ribs , Passing through the entire posterior region. The balance of each individual will be evaluated in the force platform at four different times, before, immediately after, after 24 and 48 hours after the application of the bandage, in three different tasks of postural control in the force platform, being: unipedal right, unipedal left and task Of bipedal support in the semi-tandem position. Will be performed three evaluations of 30s each, with 30s of interval between each evaluation.
  Interventions: Device: Bandage

INTERVENTIONS:
Device: Bandage — Application of Elastic Bandage Therapy by the Therapy Taping method
  Other Names: Therapy Taping; Elastic Tape; Elastic bandage; Therapeutic elastic bandage

SUMMARY:
Elastic Bandaging Therapy (BET) is a technique that consists of the application of elastic adhesive tape directed on a skin, and is used for pain reduction, improvement of flexibility, postural alignment. It is believed that it can help proprioception by increasing or reducing muscle tension by acting on motor coordination and balance. The present study aims to evaluate the effect of the application of different BET strategies on the postural balance of healthy young women through measures obtained through a proper instrument for a balance assessment, a force platform.

ELIGIBILITY:
Inclusion Criteria:

* women aged between 18 and 35 years;
* not present chronic pain defined as daily or almost daily pain during the last three months;
* not participate in rehabilitation programs.

Exclusion Criteria:

* present any type of neurological, cardiorespiratory, metabolic and / or orthopedic disease of high severity;
* vestibulopathies and labyrinthine crises;
* mental problems, attention and speech disorders;
* some other type of impediment or problem that interfered with physical and functional tests;
* Have undergone some kind of locomotor surgery;
* pregnancy;
* no participation in the three days of the research;
* lack of understanding or non-cooperation regarding research procedures and methods;
* do not volunteer.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2016-05-01 (Actual); Primary Completion 2017-02-01 (Actual); Study Completion 2017-02-01 (Actual)

PRIMARY OUTCOMES:
Changes in center of Pressure Area (COP) | Before the application of the bandage (Pre-intervention), immediately after, twenty-four hours after and forty-eight hours after the application of the bandage
  Ellipse area (95%) of the center of pressure (COP) in cm2

SECONDARY OUTCOMES:
Mean velocity in anteroposterior direction (VAP) | Before the application of the bandage (Pre-intervention), immediately after, twenty-four hours after and forty-eight hours after the application of the bandage
  Mean velocity (cm/s) of COP oscillation in the anteroposterior direction of movement
Mean velocity in the mid-lateral direction (VML) | Before the application of the bandage (Pre-intervention), immediately after, twenty-four hours after and forty-eight hours after the application of the bandage
  Mean velocity (cm/s) of COP oscillation in the mid-lateral direction of movement
Mean frequency in anteroposterior direction (FAP) | Before the application of the bandage (Pre-intervention), immediately after, twenty-four hours after and forty-eight hours after the application of the bandage
  Mean frequency (in Hz) of COP oscillation in the anteroposterior direction of movement
Mean frequency in the mid-lateral direction (FML) | Before the application of the bandage (Pre-intervention), immediately after, twenty-four hours after and forty-eight hours after the application of the bandage
  Mean frequency (in Hz) of COP oscillation in the mid-lateral direction of movement

IPD SHARING:
Plan to Share IPD: No